CLINICAL TRIAL: NCT07245758
Title: Stryker Customized Plates for Mandibular Reconstruction: A Retrospective Post Market Follow Up to Confirm Safety and Performance of Facial iD Customized Mandible Reconstruction Plates
Brief Title: Facial iD Customized Mandible Reconstruction Plates
Status: Recruiting | Type: Observational
Sponsor: Stryker Craniomaxillofacial (Industry)
Responsible Party: Sponsor
Other Study IDs: CMRP_2023_01_CIP_v 1.0
Record Dates: First submitted 2025-07-31; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Mandibular Fractures; Mandible Fracture; Mandible; Deformity; MANDIBLE; Orthognathic Surgical Procedures
Keywords: Mandibular Reconstruction; Reconstruction Plate; Orthognathic Surgery; Mandibular Reconstruction* / Methods
MeSH Terms: conditions — Mandibular Fractures; Congenital Abnormalities | interventions — Mandibular Reconstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Mandibular reconstruction — Primary or secondary reconstruction of the mandible using customized Mandible Reconstruction Plate (referred to as CMRP)

SUMMARY:
A retrospective post market follow up to confirm the safety and performance of Stryker's Customized Plates for Mandibular Reconstruction. The study is performed to confirm the product's performance and safety by systematically collecting clinical data on its use.

DETAILED DESCRIPTION:
This is a retrospective non-interventional post-market follow up aiming at confirming safety and performance of Stryker Customized Plates for Mandibular Reconstruction (CMRP) in the clinical setting. his study will include patients who have previously undergone a surgical procedure involving the Study Device, with surgical outcomes evaluated retrospectively. The Customized Mandible Recon Plate Kit is indicated for use in primary mandibular reconstruction with bone graft, temporary bridging until delayed secondary reconstruction and secondary mandibular reconstruction. Up to 3 investigational sites in US will be participating. Based on a non-inferiority study power calculation 80 subjects will be enrolled in the study. The primary outcome parameter evaluating successful reconstruction of the mandible without the need for unplanned revision surgery will be evaluated at all available follow-up timepoints of the included patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent primary or secondary mandibular reconstruction using a Stryker Facial iD CMRP implant as per routine clinical practice.
2. Patients for whom data on the primary outcome variable is available.

Exclusion Criteria:

1. Patients with active local infections at the time of surgery
2. Patients with known metal allergies and/or foreign body sensitivity at the time of surgery
3. Potentially non-compliant patients who were unwilling or incapable of following post-operative care instructions
4. Patients with inadequate bone quantity or quality necessary for plate fixation or stabilization at the time of surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will be identified as having had a surgical procedure involving the Subject Device.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of successful reconstruction of the mandible without the need for unplanned revision surgery | Data collected at a single time point per patient in the course of 16 months
  Rate of unplanned revision surgery determined by reviewing adverse events in patient medical charts after surgery. Used to document whether an unplanned revision surgery was required or not for each patient.

SECONDARY OUTCOMES:
Rate of satisfactory occlusion achieved with orthodontic treatment. | Data collected at a single time point per patient in the course of 16 months.
  Assessed by review of individual patient medical records that document the rate of satisfactory occlusion achieved with orthodontic treatment.
Infection rate | Data collected at time points from patient medical charts in the course of 16 months.
  Determined by adverse events reported from patient medical charts.
Intraoperative complications | Data collected at a single time point per patient in the course of 16 months.
  Determined by adverse events reported from patient medical charts.
Postoperative complications | Data collected at time points per patient in the course of 16 months.
  Determined by adverse events reported from patient medical charts.
Any known adverse events | Data collected at time points per patient in the course of 16 months.
  Determined by adverse events reported from patient medical charts.
Rate of plate or screw failure | Data collected at time points point per patient in the course of 16 months.
  Determined by rate of adverse events reported from patient medical charts involving plate or screw fracture.
Operating room (OR) time | Data collected at a single time point per patient in the course of 16 months.
  Time patients are operated (dd:hh)
Time to return to solid food/normal diet | Data collected at a single time point per patient in the course of 16 months.
  Time for patient to return to solid food/normal diet post operation (dd)
Hospitalization time: ICU and normal ward | Data collected at a single time point per patient in the course of 16 months.
  Time the patient was hospitalized post procedure (dd:hh)
EuroQol-5 Domain Questionnaire (if available) | Data collected at time points per patient in the course of 16 months.
  A descriptive system and a visual analogue scale (VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each with three to five levels of severity. The VAS provides a subjective rating of overall health on a scale from 0 to 100 (higher is better)).
End user questionnaire | Data collected during the course of 16 months.
  Questionnaire only for medically trained professionals on site staff using the device. Questions relate to subjective rating of ease of use by the surgeon if compared to stock plates (evaluated per treating surgeon, not per patient). Questionnaire is qualitative response regarding the ease of use of the device.
Misfit of implant | Data collected at time points per patient in the course of 16 months.
  Fit of implant Time for adaptations
Facial Appearance, Quality of Life, and Satisfaction Questionnaire (if available) | Data collected at time points per patient in the course of 16 months.
  40 independently functioning scales and checklists. Multiple independent scales, each with a 0-100 score, where higher scores indicate better outcomes. Scores are calculated by summing responses on a 4-point Likert scale (e.g., strongly disagree to strongly agree), which are then converted to the 0-100 range. Each scale measures a specific aspect of facial appearance, quality of life, or adverse effects and cannot be summed into a single total score.
12-Item Short Form Health Survey (SF-12) | Data collected at time points per patient in the course of 16 months.
  12 items grouped and scored to produce two separate summary scores: the Physical Component Summary (PCS-12) and the Mental Component Summary (MCS-12). The scale is transformed to a 0-100 range with higher scores indicating better health.
Visual Analogue Scale (VAS) Pain | Data collected at time points per patient in the course of 16 months.
  The visual analogue scale (VAS) is a psychometric response scale. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). 100-mm VAS ratings of 0 to 4 mm can be considered no pain; 5 to 44 mm, mild pain; 45 to 74 mm, moderate pain; and 75 to 100 mm, severe pain.
Ischemia time | Data collected at a single time point per patient in the course of 16 months.
  Ischemia time (dd:hh)
Frequency of Maxilla-mandibular fixation | Data collected at time points per patient in the course of 16 months.
  Number of maxillo-mandibular fixation procedures (number per patient).

OTHER OUTCOMES:
Follow-up time | Data collected at a single time point per patient in the course of 16 months.
  Post operative follow up time for patients within standard of care. Reported in patient medical charts during hospital follow up visits.
Flap used | Data collected at a single time point per patient in the course of 16 months.
  Type of flap used: vascularized fibula flap, vascularized scapula flap, vascularized iliac crest flap, avascularized fibula flap, avascularized scapula flap, avascularized iliac crest flap, others
Radiation | Data collected at time points per patient in the course of 16 months.
  Exposure of patient to radiation therapy within 12 months around the surgery date recorded in patient medical charts.
  Radiation therapy performed on the anatomical area treated with the device. Any postoperative radiation therapy recorded in patient medical charts.
Dental reconstruction in a single stage surgery | Data collected at time points per patient in the course of 16 months.
  Data for dental reconstruction collected from patient medical charts.
Sterilization method used | Data collected at a single time point per patient in the course of 16 months.
  Sterilization method used for the device.
Fixation system used | Data collected at a single time point per patient in the course of 18 months.
  System used to fix the device during the procedure. Stryker Universal Mandible System; other
  Types and number of screws
Plate types | Data collected at a single time point per patient in the course of 16 months.
  2.0 or 2.8 plates used Hemi or full reconstruction plate used
Patient age | Data collected at a single time point per patient in the course of 16 months.
  Age (years)
Gender | Data collected at a single time point per patient in the course of 16 months
  Responses: Male, Female, undifferentiated, unknown
Primary indication for the surgery / diagnosis | Data collected at a single time point per patient in the course of 16 months.
  Diagnosis collected from patient medical charts.
Surgical approach | Data collected at a single time point per patient in the course of 16 months.
  Surgical approach taken for the procedure. Including: transoral; transbuccal; submandibular; preauricular; other
Relevant Medical conditions | Data collected at time points per patient in the course of 16 months.
  Descriptive data of any underlying medical conditions and medications recorded in patient medical charts that may be related to the device or primary outcome (qualitative measure).
Primary/secondary reconstruction performed | Data collected at time points point per patient in the course of 16 months
  Type of reconstruction procedure performed (e.g. immediately or after an initial surgery).
Localization of the defect | Data collected at time points point per patient in the course of 16 months.
  Area to treated by the device: mandibular ramus; mandibular body; mandibular condyle; parasymphysis; paramedian; other
Patient height | Data collected at a single time point per patient in the course of 16 months.
  Height (cm, feet, inches)
Patient weight | Data collected at a single time point per patient in the course of 16 months.
  Weight (kg, lb)
Year smoking was stopped | Data collected at time points per patient in the course of 16 months.
  Year smoking was stopped (YYYY)
Smoking frequency | Data collected at time points per patient in the course of 16 month
  The frequency of exposure to smoking during periods of smoking (average number of cigarettes per day).
Smoking duration | Data collected at time points per patient in the course of 16 month
  Duration of smoking (pack years)
Years of active smoking | Data collected at time points per patient in the course of 16 month
  Total number of years active smoker (YY)

CONTACTS AND LOCATIONS:
Locations (1):
- Head & Neck Surgery Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] van Baar GJC, Forouzanfar T, Liberton NPTJ, Winters HAH, Leusink FKJ. Accuracy of computer-assisted surgery in mandibular reconstruction: A systematic review. Oral Oncol. 2018 Sep;84:52-60. doi: 10.1016/j.oraloncology.2018.07.004. Epub 2018 Jul 20. PMID 30115476
- [Background] Mollmann HL, Apeltrath L, Karnatz N, Wilkat M, Riedel E, Singh DD, Rana M. Comparison of the Accuracy and Clinical Parameters of Patient-Specific and Conventionally Bended Plates for Mandibular Reconstruction. Front Oncol. 2021 Nov 26;11:719028. doi: 10.3389/fonc.2021.719028. eCollection 2021. PMID 34900674
- [Background] Witjes MJH, Schepers RH, Kraeima J. Impact of 3D virtual planning on reconstruction of mandibular and maxillary surgical defects in head and neck oncology. Curr Opin Otolaryngol Head Neck Surg. 2018 Apr;26(2):108-114. doi: 10.1097/MOO.0000000000000437. PMID 29470184
- [Background] Lee ZH, Alfonso AR, Ramly EP, Kantar RS, Yu JW, Daar D, Hirsch DL, Jacobson A, Levine JP. The Latest Evolution in Virtual Surgical Planning: Customized Reconstruction Plates in Free Fibula Flap Mandibular Reconstruction. Plast Reconstr Surg. 2020 Oct;146(4):872-879. doi: 10.1097/PRS.0000000000007161. PMID 32590512
- [Background] Kakarala K, Shnayder Y, Tsue TT, Girod DA. Mandibular reconstruction. Oral Oncol. 2018 Feb;77:111-117. doi: 10.1016/j.oraloncology.2017.12.020. Epub 2018 Jan 4. PMID 29362116